CLINICAL TRIAL: NCT06936085
Title: Forensic Case and Forensic Evidence Management Training: Paramedic Student Example
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Yeliz Sapulu Alakan, Lecturer, Uludag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: forensic cases
Record Dates: First submitted 2025-04-06; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Training Effectiveness; Training; Student Education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Other): The data for the study were collected between May 2024 and June 2024. The students included in the study were given a data collection form before and after the training.
  The Crime Scene Forensic Evidence Management training, which included theoretical knowledge and the presentation of sample cases, was completed for 144 volunteer participants. The content of the training includes topics such as forensic incidents, evidence, crime scene management, and evidence management, as well as the roles and responsibilities of paramedics in forensic cases such as injuries, violence, abuse, sexual assault, and suicide. Training was given to 4 groups of 35-37 students in each group in the classroom environment in two class hours (30+ 30 minutes + 1 break). Trainings were given by a single lecturer to avoid bias and ensure standardization.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — The Crime Scene Forensic Evidence Management training, which included theoretical knowledge and the presentation of sample cases, was completed for 144 volunteer participants. The content of the training includes topics such as forensic incidents, evidence, crime scene management, and evidence management, as well as the roles and responsibilities of paramedics in forensic cases such as injuries, violence, abuse, sexual assault, and suicide. Training was given to 4 groups of 35-37 students in each group in the classroom environment in two class hours (30+ 30 minutes + 1 break). Trainings were given by a single lecturer to avoid bias and ensure standardization.

SUMMARY:
This study aimed to provide forensic case and evidence management training to paramedic students and to evaluate the effect of the training on the knowledge level of the students.

ELIGIBILITY:
Inclusion Criteria:

* Paramedic students studying in the 1st and 2nd grades of the First and Emergency Aid Programme who volunteered to participate in the study.

Exclusion Criteria:

* Paramedic students who are not studying in the First and Emergency Aid Programme and who did not volunteer for the research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
questionnaire | The evaluation was performed on the same day before and after the training.
  to evaluate the effect of the training on the knowledge level of the students.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Information is planned to be shared at the publication stage.